CLINICAL TRIAL: NCT02174549
Title: Phase I Dose-Escalating Study of Combining Intravenous Tirapazamine and Transarterial Embolization (TAE) in Liver Cancer
Brief Title: Dose-defining Study of Tirapazamine Combined With Embolization in Liver Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teclison Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT001
Record Dates: First submitted 2014-06-10; First posted 2014-06-25 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Gastrointestinal Cancer Metastatic; Neuroendocrine Tumors
Keywords: Hypoxia; Embolization; Tirapazamine
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neuroendocrine Tumors; Hypoxia | interventions — Tirapazamine; Ethiodized Oil

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation 3+3 design completed; now only for expansion cohort in neuroendocrine tumor.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tirapazamine (Experimental): Intra-arterial administration with tirapazamine before embolization to evaluate the response in metastatic liver lesions of NET
  Interventions: Drug: Tirapazamine; Procedure: Conventional Transarterial Embolization (TAE)

INTERVENTIONS:
Drug: Tirapazamine — Intra-arterial injection into the tumor feeding artery
Procedure: Conventional Transarterial Embolization (TAE) — Lipiodol and Gelfoam used to embolize tumor vessels and induce tumor hypoxia
  Other Names: TAE conducted with Lipiodol and Surgifoam as the embolizing agents.

SUMMARY:
This phase 1 study is to determine the optimal dose and tolerability of a hypoxia-activating agent, tirapazamine, when it is combined with embolization in liver cancer. Liver cancer patients who are Child-Pugh score A, suitable for embolization with tumor no more than 4 nodules are eligible. Tirapazamine will be given by intra-arterial injection before embolization. Treatment effect is evaluated by MRI based on mRECIST criteria. Repeat treatment is necessary only if disease progression. Dose escalation cohort has been completed. Expansion cohort is open for metastatic liver dominant neuroendocrine tumor.

DETAILED DESCRIPTION:
The study is a 3+3 design for dose escalation. Each cohort will have 3-6 patients based on tolerability. Patients will receive escalated doses of tirapazamine until maximally tolerated dose. Embolization is performed per standard practice using Lipiodol and Gelfoam under X-ray guidance. Once a suitable dose is determined, an expansion cohort of 15 patients will be treated with the recommended phase 2 dose to determine preliminary efficacy. Expansion cohorts include (1) hepatocellular carcinoma, (2) metastatic solid tumors with liver metastasis, and (3) neuroendocrine tumor. Adverse events are evaluated by CTCAE vs. 5.0 and efficacy is evaluated by MRI using modified RECIST criteria and RECIST criteria.

The dose escalation part has been completed. Only the third cohort or neuroendocrine tumor remains active for future patient enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with well-differentiated NET and liver-dominant metastatic disease with intrahepatic disease progression, regardless of primary tumor origin or tumor functional status. Patients may have extrahepatic lesions as long as the majority of the disease burden is intrahepatic.
2. No limitation in hepatic lesion tumor size or number but the total volume of liver tumors cannot exceed 50% of the liver volume.
3. Patients are allowed to have prior US Food and Drug Administration (FDA)-approved treatments, including systemic therapies, surgery, ablation, or transarterial therapies for the metastatic NET.
4. Age 20 or higher, ECOG functional status 0-1, and with no known major cardiac, pulmonary, or renal dysfunction.
5. Are candidates for TAE or TACE and without portal vein occlusion per treating interventional radiologists.
6. ANC no less than 1000 /μL. Hemoglobin ≥ 9 gm/dL. Platelets no less than 50,000 /μL. Creatinine no more than 2.0 mg/dL. AST, ALT no more than 5X upper limit of normal. Bilirubin no more than 2.5 mg/dl. PT prolongation ≤ 4 sec above upper limit of normal.
7. Woman of child-bearing potential (WOCBP) should use highly effective contraception during trial participation and for 6 months after the last dose of tirapazamine and men who are partners with WOCBP should use highly effective contraception, including barrier contraception, during trial participation and for 3 months after the last dose of tirapazamine.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-09; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response rate (ORR) by RECIST | 2 years
  Overall Response Rate by RECIST criteria

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  Overall Response Rate by mRECIST criteria
Duration of Response | 2 years
  Duration of Response by RECIST and mRECIST

OTHER OUTCOMES:
Response Rate in TATE-treated target lesions | 2 years
  by mRECIST and RECIST
Progressive Free Survival | 2 years
  by RECIST and mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soulen, MD, Principal Investigator — Univ. of Pennsylvania
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abi-Jaoudeh N, Dayyani F, Chen PJ, Fernando D, Fidelman N, Javan H, Liang PC, Hwang JI, Imagawa DK. Phase I Trial on Arterial Embolization with Hypoxia Activated Tirapazamine for Unresectable Hepatocellular Carcinoma. J Hepatocell Carcinoma. 2021 May 17;8:421-434. doi: 10.2147/JHC.S304275. eCollection 2021. PMID 34041204
- See also: Phase 1 dose escalation result in Hepatocellular carcinoma — https://pubmed.ncbi.nlm.nih.gov/34041204/